CLINICAL TRIAL: NCT02494518
Title: Forced Aerobic Exercise for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Susan Linder, Research Physical Therapist, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-402
Record Dates: First submitted 2015-07-06; First posted 2015-07-10 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2018-12

CONDITIONS: Stroke
Keywords: stroke; aerobic exercise; forced exercise; repetitive task practice; arm function; upper extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Forced Exercise & Upper Extremity Repetitive Task Practice (Active Comparator): Participants will perform the following:
  1. 45 minutes of cycling on a recumbent stationary bike with a specialized motor that forces the individual to cycle approximately 30-35% faster than your self-selected speed
  2. 45 minutes of upper extremity repetitive arm exercises
  Interventions: Behavioral: Forced Exercise & Upper Extremity Repetitive Task Practice
- Voluntary Exercise & Upper Extremity Repetitive Task Practice (Active Comparator): Participants will perform the following:
  1. 45 minutes of cycling on a recumbent stationary bike at your self-selected speed
  2. 45 minutes of upper extremity repetitive arm exercises
  Interventions: Behavioral: Voluntary Exercise & Upper Extremity Repetitive Task Practice
- Stroke Education & Upper Extremity Repetitive Task Practice (Active Comparator): Participants will perform the following:
  1. 45 minutes of stroke education
  2. 45 minutes of upper extremity repetitive arm exercises
  Interventions: Behavioral: Stroke Education & Upper Extremity Repetitive Task Practice

INTERVENTIONS:
Behavioral: Forced Exercise & Upper Extremity Repetitive Task Practice
  Arms: Forced Exercise & Upper Extremity Repetitive Task Practice
Behavioral: Voluntary Exercise & Upper Extremity Repetitive Task Practice
  Arms: Voluntary Exercise & Upper Extremity Repetitive Task Practice
Behavioral: Stroke Education & Upper Extremity Repetitive Task Practice
  Arms: Stroke Education & Upper Extremity Repetitive Task Practice

SUMMARY:
The purpose of the study is to determine if performing different types of aerobic exercise (cycling) before upper extremity exercises will help to improve outcomes after stroke.

DETAILED DESCRIPTION:
The goal of this study is to determine the potential for forced aerobic exercise to augment the recovery of motor function in individuals with stroke. Current approaches to stroke rehabilitation involve intensive, therapist-directed task practice that is both expensive and in some cases, ineffective in fostering functional neuromotor recovery. The identification of a safe, cost-effective approach, such as forced aerobic exercise, to augment the recovery of function achieved through task practice while simultaneously decreasing the cardiovascular risk factors prevalent in stroke survivors would be significant to rehabilitation and stroke communities.

Animal studies along with preliminary human data indicate a specific type of aerobic exercise (AE), forced aerobic exercise (FE), may be ideal in facilitating motor recovery associated with repetitive task practice (RTP). The hypothesis is that that deficits in afferent input and motor cortical output following stroke prevents patients from achieving and maintaining an exercise intensity that is sufficient for facilitating motor recovery; therefore, FE is needed to augment their voluntary efforts and achieve greater gains in recovery. In previous research, a safe lower extremity FE intervention was initially applied to individuals with Parkinson's disease and subsequently to individuals with stroke. Preliminary results indicate that those completing an 8-week FE intervention paired with an abbreviated session of RTP exhibited significantly greater improvement in Fugl-Meyer scores at end of treatment despite completing 40% fewer RTP repetitions, compared to those receiving voluntary-rate aerobic exercise (VE) and RTP and time-matched RTP only. Improvements in cardiovascular fitness and lower extremity motor function were also evident in both groups that engaged in aerobic exercise (FE and VE). Positive results from a preliminary trial indicate safety, feasibility, and initial efficacy of combining two modes of aerobic exercise training with RTP provide rationale for a systematic and larger scale trial to determine the precise role of aerobic exercise, forced and voluntary, in facilitating motor recovery following stroke.

For this study, 30 individuals with chronic stroke will be randomized into one of the following groups: FE = RTP, VE + RTP or patient education and RTP. All three groups will receive an identical dose of contact time over 8 weeks (3X per week). An intervention group receiving a 45-minute session of patient education paired with RTP will serve as the non-exercise control. Clinical and biomechanical outcomes measuring change in upper extremity motor function, lower extremity motor function, and cardiovascular fitness will provide the most complete picture, to date, on the potential neurologic effects of AE (forced and voluntary) on motor recovery and brain function in humans with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* At least 6 months post diagnosis of single ischemic stroke, confirmed with neuroimaging
* Fugl-Meyer Motor Score 19-55 in involved upper extremity
* Approval from patient's physician
* Age between 18 and 85 years

Exclusion Criteria:

* Hospitalization for myocardial infarction, congestive heart failure, or heart surgery (CABG or valve replacement) within 3 months of study enrollment
* Serious cardiac arrhythmia
* Other serious heart and lung conditions (i.e.cardiomyopathy, aortic stenosis, cardiac pacemaker, pulmonary embolus)
* Other medical or musculoskeletal contraindication to exercise
* Significant cognitive impairment (unable to follow 1-2 step commands) or major psychiatric disorder (major depression, generalized anxiety) that will cause difficulty in study participation
* Anti-spasticity injection (botox) in upper extremity within 3 months of study enrollment
* Pregnancy
* Unstable blood pressure at rest or with exercise

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-07; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Linder, PT, DPT, NCS, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Linder SM, Davidson S, Rosenfeldt A, Lee J, Koop MM, Bethoux F, Alberts JL. Forced and Voluntary Aerobic Cycling Interventions Improve Walking Capacity in Individuals With Chronic Stroke. Arch Phys Med Rehabil. 2021 Jan;102(1):1-8. doi: 10.1016/j.apmr.2020.08.006. Epub 2020 Sep 9. PMID 32918907
- [Derived] Linder SM, Davidson S, Rosenfeldt A, Penko A, Lee J, Koop MM, Phelan D, Alberts JL. Predictors of Improved Aerobic Capacity in Individuals With Chronic Stroke Participating in Cycling Interventions. Arch Phys Med Rehabil. 2020 Apr;101(4):717-721. doi: 10.1016/j.apmr.2019.10.187. Epub 2019 Nov 25. PMID 31778659
- [Derived] Rosenfeldt AB, Linder SM, Davidson S, Clark C, Zimmerman NM, Lee JJ, Alberts JL. Combined Aerobic Exercise and Task Practice Improve Health-Related Quality of Life Poststroke: A Preliminary Analysis. Arch Phys Med Rehabil. 2019 May;100(5):923-930. doi: 10.1016/j.apmr.2018.11.011. Epub 2018 Dec 10. PMID 30543801

RESULTS

PARTICIPANT FLOW:
Groups:
- Forced Exercise & Upper Extremity Repetitive Task Practice: Participants will perform the following:
  1. 45 minutes of cycling on a recumbent stationary bike with a specialized motor that forces the individual to cycle approximately 30-35% faster than your self-selected speed
  2. 45 minutes of upper extremity repetitive arm exercises
  Forced Exercise & Upper Extremity Repetitive Task Practice
- Voluntary Exercise & Upper Extremity Repetitive Task Practice: Participants will perform the following:
  1. 45 minutes of cycling on a recumbent stationary bike at your self-selected speed
  2. 45 minutes of upper extremity repetitive arm exercises
  Voluntary Exercise & Upper Extremity Repetitive Task Practice
- Stroke Education & Upper Extremity Repetitive Task Practice: Participants will perform the following:
  1. 45 minutes of stroke education
  2. 45 minutes of upper extremity repetitive arm exercises
  Stroke Education & Upper Extremity Repetitive Task Practice
Period: Overall Study
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Started | 11 | 12 | 11
Completed | 10 | 10 | 8
Not Completed | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice | Total
Number analyzed (Participants) | 11 | 12 | 11 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 6 | 21
  >=65 years | 3 | 5 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.91 (10.69) | 59.33 (13.84) | 60.45 (11.25) | 58.26 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 13
  Male | 7 | 6 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 10 | 11 | 10 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 6 | 15
  White | 3 | 7 | 3 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 11 | 34
Fugl-Meyer Assessment [Mean (Standard Deviation); unit: units on a scale] — Motor test to assess arm impairment. Scores range from 0-66 and higher scores represent less impairment.
  units on a scale | 35.73 (8.71) | 35.92 (10.11) | 32.09 (7.44) | 34.62 (8.77)
Wolf Motor Function Test [Mean (Standard Deviation); unit: units on a scale] — Motor test to assess arm function. The reported data is the total Functional Ability Score. Scores range from 0-75 and higher scores represent improved function.
  units on a scale | 55.09 (12.19) | 52.83 (9.49) | 51.91 (8.79) | 53.26 (10.02)
Stroke Impact Scale [Mean (Standard Deviation); unit: units on a scale] — Quality of life questionnaire. The reported data is the normalized Hand Function score. Scores range from 0-100, with higher scores indicating better perceived hand function.
  units on a scale | 53.64 (23.46) | 51.67 (18.13) | 54.09 (20.23) | 53.09 (20.04)
Metabolic Stress Test [Mean (Standard Deviation); unit: mL/kg/min] — Cycling test to measure cardiovascular fitness. The data reported is VO2peak. Higher scores indicate higher aerobic capacities.
  mL/kg/min | 15.23 (3.84) | 16.72 (4.06) | 14.58 (3.48) | 15.54 (3.81)

OUTCOME MEASURES:

1. Primary Outcome: Fugl Meyer Assessment
Description: Motor test to assess arm impairment. The reported data is the change in total score. Score range from 0-66 and higher scores represent less impairment.
Time Frame: Change from baseline to midpoint (4 weeks into treatment), at end of 8 week intervention, and 4 weeks after the intervention ends
Population: One individual in FE+RTP completed EOT but was lost to follow-up and did not complete EOT+4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Number analyzed (Participants) | 10 | 10 | 8
units on a scale
  Baseline to Midpoint | 6.90 (5.55) | 4.00 (3.27) | 6.25 (3.65)
  Baseline to EOT | 10.10 (5.32) | 6.50 (3.47) | 8.88 (4.76)
  Baseline to EOT+4: number analyzed (Participants) | 9 | 10 | 8
  Baseline to EOT+4 | 11.11 (5.69) | 7.10 (4.51) | 9.25 (5.75)

2. Primary Outcome: Wolf Motor Function Test
Description: Motor test to assess arm function. The reported data is the change in total Functional Ability Score. Scores range from 0-75 and higher scores represent improved function.
Time Frame: Change from baseline to end of 8 week intervention, and 4 weeks after the intervention ends
Population: One individual in FE+RTP completed EOT but was lost to follow-up and did not complete EOT+4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Number analyzed (Participants) | 10 | 10 | 8
units on a scale
  Baseline to EOT | 7.80 (6.09) | 6.40 (3.17) | 10.50 (6.87)
  Baseline to EOT+4: number analyzed (Participants) | 9 | 10 | 8
  Baseline to EOT+4 | 9.22 (6.67) | 9.60 (2.59) | 10.88 (6.77)

3. Primary Outcome: Stroke Impact Scale
Description: Quality of life questionnaire. The reported data is the normalized Hand Function score. Scores range from 0-100, with higher scores indicating better perceived hand function.
Time Frame: Change from baseline to end of 8 week intervention, and 4 weeks after the intervention ends
Population: One individual in FE+RTP completed EOT but was lost to follow-up and did not complete EOT+4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Number analyzed (Participants) | 10 | 10 | 8
units on a scale
  Baseline to EOT | 15.00 (11.55) | 14.50 (14.03) | 9.38 (12.08)
  Baseline to EOT+4: number analyzed (Participants) | 9 | 10 | 8
  Baseline to EOT+4 | 19.44 (12.10) | 14.00 (20.25) | 21.25 (19.04)

4. Primary Outcome: Metabolic Stress Test
Description: Cycling test to measure cardiovascular fitness. The data reported is the change in VO2peak. Higher scores indicate higher aerobic capacities.
Time Frame: Change from baseline to follow up assessments at end of 8 week intervention
Measure: Mean (Standard Error); unit: mL/kg/min
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Number analyzed (Participants) | 10 | 9 | 8
mL/kg/min | 0.02 (1.35) | 1.09 (1.70) | 0.40 (0.70)

5. Secondary Outcome: Action Research Arm Test
Description: Motor test to assess arm function. The reported data is change in total score. Scores range from 0-57, and higher scores indicate better function.
Time Frame: Change from baseline to end of 8 week intervention, and 4 weeks after the intervention ends
Population: One individual in FE+RTP completed EOT but was lost to follow-up and did not complete EOT+4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Number analyzed (Participants) | 10 | 10 | 8
units on a scale
  Baseline to EOT | 8.60 (6.24) | 6.30 (4.83) | 6.38 (4.96)
  Baseline to EOT+4: number analyzed (Participants) | 9 | 10 | 8
  Baseline to EOT+4 | 8.56 (4.98) | 7.50 (5.50) | 7.13 (4.52)

6. Secondary Outcome: Center for Epidemiological Studies-Depression
Description: Depression questionnaire. The reported data is change in total score. Scores range from 0-60, and lower scores indicate decreased risk of depression.
Time Frame: Change from baseline to end of 8 week intervention, and 4 weeks after the intervention ends
Population: One individual in FE+RTP completed EOT but was lost to follow-up and did not complete EOT+4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Number analyzed (Participants) | 10 | 10 | 8
units on a scale
  Baseline to EOT | -5.20 (7.44) | -0.30 (8.31) | -2.00 (5.53)
  Baseline to EOT+4: number analyzed (Participants) | 9 | 10 | 8
  Baseline to EOT+4 | -3.67 (6.63) | -2.60 (5.46) | -3.75 (7.21)

7. Secondary Outcome: Processing Speed Test
Description: Matching letters and symbols to test cognition. The reported data is change in total number correct.
Time Frame: Change from baseline to end of 8 week intervention, and 4 weeks after the intervention ends
Population: One individual in FE+RTP completed EOT but was lost to follow-up and did not complete EOT+4
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Number analyzed (Participants) | 10 | 10 | 8
number correct
  Baseline to EOT | 0.90 (4.68) | 1.88 (4.22) | 2.71 (6.32)
  Baseline to EOT+4: number analyzed (Participants) | 9 | 10 | 8
  Baseline to EOT+4 | 2.89 (7.52) | 3.25 (5.15) | 6.38 (10.27)

8. Secondary Outcome: Nine Hole Peg Test
Description: Transferring pegs into a fitted hole to measure hand function. The reported data is change in average time to complete.
Time Frame: Change from baseline to end of 8 week intervention, and 4 weeks after the intervention ends
Population: One individual in FE+RTP completed EOT but was lost to follow-up and did not complete EOT+4. One individual in VE+RTP did not complete the NHPT at EOT+4.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Number analyzed (Participants) | 10 | 10 | 8
seconds
  Baseline to EOT | -8.07 (15.71) | -16.15 (45.64) | -19.35 (21.51)
  Baseline to EOT+4: number analyzed (Participants) | 9 | 9 | 8
  Baseline to EOT+4 | -8.10 (10.58) | -7.81 (34.89) | -29.15 (32.75)

9. Secondary Outcome: Six Minute Walk Test
Description: Distance walked in 6 minutes to measure cardiovascular fitness. The reported data is change in total distance traveled.
Time Frame: Change from baseline to end of 8 week intervention, and 4 weeks after the intervention ends
Population: Two individuals in FE+RTP did not complete this assessment at EOT+4
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
Number analyzed (Participants) | 10 | 10 | 8
feet
  Baseline to EOT | 133.20 (107.78) | 188.70 (155.22) | -21.75 (111.76)
  Baseline to EOT+4: number analyzed (Participants) | 8 | 10 | 8
  Baseline to EOT+4 | 78.50 (224.32) | 127.70 (190.05) | 78.88 (202.38)

ADVERSE EVENTS:
Time Frame: 12 weeks from baseline assessment
Arm/Group | Forced Exercise & Upper Extremity Repetitive Task Practice | Voluntary Exercise & Upper Extremity Repetitive Task Practice | Stroke Education & Upper Extremity Repetitive Task Practice
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 1/11
Other Adverse Events (participants affected / at risk) | 1/11 | 0/12 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forced Exercise & Upper Extremity Repetitive Task Practice (N=11) | Voluntary Exercise & Upper Extremity Repetitive Task Practice (N=12) | Stroke Education & Upper Extremity Repetitive Task Practice (N=11)
Fall (General disorders) | 0 (0) | 0 (0) | 1 (1) — One participant fell during 6MWT administration, resulting in superficial injuries that did not require follow up care.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forced Exercise & Upper Extremity Repetitive Task Practice (N=11) | Voluntary Exercise & Upper Extremity Repetitive Task Practice (N=12) | Stroke Education & Upper Extremity Repetitive Task Practice (N=11)
Skin Integrity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — One participant developed a blister after forced exercise. The blister was monitored and did not require follow up care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-04-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT02494518/Prot_SAP_000.pdf